CLINICAL TRIAL: NCT07155720
Title: Effects of Kinesio Taping on Premenstrual Syndrome, Happiness, and Quality of Life
Brief Title: Effects of Kinesio Taping on Premenstrual Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yağmur SÜRMELİ (Other)
Responsible Party: Sponsor-Investigator, Yağmur SÜRMELİ, Asst. Prof, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/009
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Over 18 Years Old
Keywords: kinesio-tape; kinesio-taping; nursing; happiness; quality of life
MeSH Terms: interventions — Methods; Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (Experimental): Kinesio tape will be applied with 100% tension.
  Interventions: Other: Intervention (Kinesio Taping) group
- Sham Taping (Placebo Comparator): Kinesio tape will be applied without tension.
  Interventions: Other: Intervention (Kinesio Taping) group

INTERVENTIONS:
Other: Intervention (Kinesio Taping) group — No studies have been found in the literature examining whether kinesio taping increases happiness in women with PMS.

SUMMARY:
This randomized, single-blind study aimed to evaluate the effects of kinesio taping on PMS symptoms, happiness, and quality of life.

The primary question(s) it aimed to answer were:

Is there a significant difference in premenstrual symptoms, happiness, and quality of life between the kinesio taping intervention group and the sham taping placebo group?

DETAILED DESCRIPTION:
The population of this study will consist of first-year female students studying in the health department at a university in the Mediterranean region between October 2025 and January 2026. The study sample will consist of women who meet the inclusion criteria and volunteer. The sample size was determined by the statistician using power analysis using the G*Power 3.1.9.4 package program. Since no studies in the literature have been found evaluating kinesio taping applied to students experiencing PMS together with the Premenstrual Syndrome Scale, the Oxford Happiness Scale, or the Premenstrual Syndrome-Specific Quality of Life Scale, Cohen's effect size values were used in the calculations. Accordingly, if an effect size was taken as 0.25, a type I error level of 0.05, a statistical power of 0.80, and a correlation coefficient between repeated measurements of 0.5, a total of 28 participants was deemed sufficient, with a minimum of 14 participants for each group. However, to prevent potential sample losses from impacting statistical power, a 25% attrition margin was anticipated, and the study was planned to include a minimum of 42 students (21 intervention, 21 placebo). Participants will be randomly selected from individuals diagnosed with PMS who meet the study criteria and divided into two groups: the intervention group (n=21) and the placebo group (n=21). Therefore, the study is planned to include a total of 42 participants.

Study participants will be assigned to intervention and placebo groups using the randomization method (https://www.randomizer.org). Data will be uploaded to the program by assigning codes to the intervention and placebo groups. Therefore, the study will also be blinded for statistical analysis and reporting. Data will be collected using the Premenstrual Syndrome Scale, the Oxford Happiness Scale, or the Premenstrual Syndrome-Specific Quality of Life Scale.

Implementation Procedure: Researcher Lecturer Yağmur Sürmeli (Y.S.) has received the internationally recognized "Kinesiology Taping Practitioner Training Certificate," which will ensure the effectiveness and efficiency of the implementation plan. Before starting the interventions, students will be provided with detailed information about the study; the researchers will assess the inclusion and exclusion criteria of students who agree to participate and sign the "Voluntary Consent Form." Before starting the kinesiology taping intervention, participants in both groups will be administered a "Descriptive Characteristics Information Form," the "Premenstrual Syndrome Scale," the Oxford Happiness Scale, and the "Premenstrual Syndrome-Specific Quality of Life Scale." Student privacy will be protected throughout the intervention, and they will be asked not to remove the tapes. Students will be instructed on how to remove the tapes and whether they should be removed before the next intervention.

Intervention Group: Students in this group will receive 100% cotton, latex-free, 5 cm x 0.5 cm original brand Kinesio Tex Gold™® kinesio tape. Application will begin one week before the estimated date of menstruation, which is when PMS symptoms are most likely to be intense. The tape will be removed on the third day after application, and a one-day break will be taken. Then, taping will be repeated in the same areas with the same tension. The application will end on the fourth day of menstruation. Kinesio taping will begin again one week before the estimated start of the next menstrual period, and the application will be repeated using the same technique as the previous month. Before each application, the skin to which the tapes will be applied will be wiped with a dry napkin. The tapes will be applied in a cross shape with 100% tension over the sacrum and in a star shape with 25-50% tension just below the clavicle. Students will complete the Premenstrual Syndrome Scale, the Oxford Happiness Scale Short Form, and the Premenstrual Syndrome-Specific Quality of Life Scale before taping, on the 4th day of their first and second menstrual periods, and on the 4th day of their third menstrual period (when the procedure is not performed).

Placebo Group: Women in this group will receive sham taping (tension-free kinesio taping). The quality of the kinesio taping will be the same as that used in the intervention group. Students will complete the Premenstrual Syndrome Scale, the Oxford Happiness Scale Short Form, and the Premenstrual Syndrome-Specific Quality of Life Scale before taping, on the 4th day of their first and second menstrual periods, and on the 4th day of their third menstrual period (when the procedure is not performed).

Statistics Statistical analysis of the data will be performed using the IBM SPSS Statistics 24.0 (IBM SPSS Statistics for Windows, Version 24.0. Armonk, NY) program. Percentage, arithmetic mean and standard deviation will be calculated in the analysis of the data. In comparing the data between two groups, Independent Two Samples t-Test (if distribution is normal) or Mann-Whitney U Test (if distribution is not normal) will be performed for continuous variables, Chi-Square Test (if data is large enough) or Fisher's Exact Test (if sample is small) will be performed for categorical variables. Repeated Measures Analysis of Variance (ANOVA), if assumptions cannot be met, non-parametric tests such as Friedman Test will be used. Bonferroni correction will be applied for interactions. In all analyses, p<0.05 will be accepted as the statistical significance level.

Ethical Aspects of the Research Ethics committee and institutional approvals will be obtained for the study. The research will be conducted in accordance with the rules of the Declaration of Helsinki (World Medical Association, 2013). All women participating in the study will be informed and their written and verbal consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Scoring at least 110 on the Premenstrual Syndrome Scale
* Having regular menstrual cycles between 28 and 35 days
* Not having any psychiatric diagnoses and not using psychiatric medications
* Not having any serious chronic diseases (e.g., diabetes, thyroid disease, cardiovascular disease)
* Being willing to participate in the study and open to communication
* Not using oral contraceptives

Exclusion Criteria:

* Having been diagnosed with an allergic skin disease
* Being pregnant
* Having a history of allergy to kinesio tape
* Having a diagnosed psychiatric disorder
* Regularly using kinesio tape
* Having serious chronic illnesses
* Student groups taught by the practitioner and the researcher
* Voluntarily withdrawing from the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women experiencing PMS
Enrollment: 42 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale | 12 weeks
  The Premenstrual Syndrome Scale was developed by Gençdoğan in 2006 to determine premenstrual symptoms. It is a five-point Liker-type scale consisting of 44 items and 9 subscales (pain, bloating, cough, anger, anxiety, depressive affect, depressive thoughts, and sleep). The lowest score on the scale is 44, and the highest is 220. The score characteristics on the scale are the increase in the intensity of PMS indicators. A minimum total score of 110 points on the PMS is classified as PMS positive. The Cronbach's α value of the scale is 0.75.

SECONDARY OUTCOMES:
Oxford Happiness Scale Short Form | 12 weeks
  Developed by Hills and Argyle (2002) and adapted into Turkish by Doğan and Akıncı-Çötok (2011), the scale is a 5-point Likert-type scale with 7 items. As the score obtained from the scale increases, the happiness level of the individual increases. The Cronbach's α value for the scale was found to be 0.74.
Premenstrual Syndrome-Specific Quality of Life Scale | 12 weeks
  The Premenstrual Syndrome-Specific Quality of Life Scale was developed by Hadavi-Bavili and İlçioğlu in 2024. The scale consists of three subscales: physical (first 11 items), emotional (items 12-18), and social (items 19-22). All items on the scale are reverse-coded. The minimum score is 22, and the maximum score is 110. Cronbach's α for the physical subscale of the scale was 0.868, for the emotional subscale was 0.846, and for the social subscale was 0.676. The scale's Cronbach's α was found to be 0.90. As the score on the scale increases, so does the quality of life.

IPD SHARING:
Plan to Share IPD: No